CLINICAL TRIAL: NCT00158600
Title: Randomized, Double-Blind, Placebo-Controlled Study of the Safety, Efficacy and Pharmacokinetics of Myozyme in Patients With Late-Onset Pompe Disease.
Brief Title: A Placebo-Controlled Study of Safety and Effectiveness of Myozyme (Alglucosidase Alfa) in Patients With Late-Onset Pompe Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AGLU02704; 2005-002759-42 (EudraCT Number)
Expanded Access: NCT00520143 (Approved for marketing)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2010-07-23 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Pompe Disease (Late-onset); Glycogen Storage Disease Type II (GSD-II); Acid Maltase Deficiency Disease; Glycogenosis 2
Keywords: Glycogen Storage Disease Type II; GSD-II; Pompe Disease
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — GAA protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- alglucosidase alfa (Active Comparator): Intravenous (IV) infusions of alglucosidase alfa at 20 milligrams (mg)/kilogram (kg) of body weight every other week (qow) for 78 weeks.
  Interventions: Biological: alglucosidase alfa
- Placebo (Placebo Comparator): Intravenous (IV) infusions of placebo every other week (qow) for 78 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: alglucosidase alfa — IV infusion of 20mg/kg; qow for 78 weeks.
  Other Names: Myozyme; Lumizyme
  Arms: alglucosidase alfa
Drug: Placebo — Placebo Comparator; qow for 78 weeks.
  Arms: Placebo

SUMMARY:
Pompe disease (also known as glycogen storage disease Type II) is caused by a deficiency of a critical enzyme in the body called acid alpha-glucosidase (GAA). Normally, GAA is used by the body's cells to break down glycogen (a stored form of sugar) within specialized structures called lysosomes. In patients with Pompe disease, an excessive amount of glycogen accumulates and is stored in various tissues, especially heart and skeletal muscle, which prevents their normal function. The overall objective is to evaluate the safety, efficacy, and pharmacokinetics (PK) of alglucosidase alfa treatment in patients with late-onset Pompe disease as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patient must provide signed, informed consent prior to performing any study-related procedures.
* Patient must have a diagnosis of Pompe disease based on deficient endogenous GAA activity in cultured skin fibroblasts of less than or equal to 40% of the normal mean of the testing laboratory and 2 confirmed GAA gene mutations;
* Patient must be greater than or equal to 8 years of age at the time of enrollment;
* Patient must be able to ambulate 40 meters (approximately 130 feet) in 6 minutes on each test performed on two consecutive days (use of assistive devices such as a walker, cane, or crutches, is permitted);
* Patient must have an FVC of greater than or equal to 30% and < 80% predicted in the upright position;
* Patient must have a postural drop in FVC (liters) of at least 10% from the upright to the supine position;
* Patient must have proximal muscle weakness in the lower limbs based on unilateral QMT of the knee extensors defined as < 80% of the predicted value based on age, gender and body size
* Patient must be able to tolerate pulmonary function testing (PFT) and muscle testing in the supine position;
* Patient must have testable muscle in bilateral knee flexors and knee extensors, and testable muscle in bilateral elbow flexors and elbow extensors;
* Patient must be able to provide reproducible muscle and pulmonary function test results;
* Patient (and patient's legal guardian if patient is < 18 years of age) must have the ability to comply with the clinical protocol;
* A female patient of childbearing potential must have a negative pregnancy test (urine) at Baseline. Note: All female patients of childbearing potential and sexually mature males must use a medically accepted method of contraception throughout the study.

Exclusion Criteria:

* Patient requires the use of invasive ventilatory support;
* Patient requires the use of noninvasive ventilatory support while awake and in an upright position;
* Patient has received enzyme replacement therapy with GAA from any source;
* Patient has used an investigational product within 30 days prior to study enrollment, or is currently enrolled in another study which involves clinical evaluations, unless prior approval is given by Genzyme;
* Patient has a major congenital anomaly, medical condition, serious intercurrent illness, or other extenuating circumstance that, in the opinion of the investigator, may significantly interfere with study compliance, including all prescribed evaluations and follow-up activities;

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2005-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (8):
- United States (5):
  - Tower Hematology Oncology Medical Group, Beverly Hills, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Washington University Medical Center, St Louis, Missouri
  - Mount Sinai School of Medicine, New York, New York
  - University of Pittsburgh, Dept. of Neurology, Pittsburgh, Pennsylvania
- Groupe Hospitalier Pitie-Salpetriere, Paris, France
- Netherlands (2):
  - Sophia Children's Hospital, Erasmus MC, Rotterdam
  - Erasmus Medical Centre Rotterdam, Rotterdam

REFERENCES:
- [Derived] Forsha D, Li JS, Smith PB, van der Ploeg AT, Kishnani P, Pasquali SK; Late-Onset Treatment Study Investigators. Cardiovascular abnormalities in late-onset Pompe disease and response to enzyme replacement therapy. Genet Med. 2011 Jul;13(7):625-31. doi: 10.1097/GIM.0b013e3182142966. PMID 21543987
- [Derived] van der Ploeg AT, Clemens PR, Corzo D, Escolar DM, Florence J, Groeneveld GJ, Herson S, Kishnani PS, Laforet P, Lake SL, Lange DJ, Leshner RT, Mayhew JE, Morgan C, Nozaki K, Park DJ, Pestronk A, Rosenbloom B, Skrinar A, van Capelle CI, van der Beek NA, Wasserstein M, Zivkovic SA. A randomized study of alglucosidase alfa in late-onset Pompe's disease. N Engl J Med. 2010 Apr 15;362(15):1396-406. doi: 10.1056/NEJMoa0909859. PMID 20393176

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One hundred patients screened and 90 enrolled.
Period: Overall Study
Arm/Group | Alglucosidase Alfa | Placebo
Started | 60 | 30
Completed | 55 | 26
Not Completed | 5 | 4
Not completed — unable to commit time to study | 0 | 1
Not completed — Adverse Event | 2 | 1
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alglucosidase Alfa | Placebo | Total
Number analyzed (Participants) | 60 | 30 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at First Infusion
  years | 45.3 (12.37) | 42.6 (11.63) | 44.4 (12.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 19 | 45
  Male | 34 | 11 | 45
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 1 | 1 | 2
  Asian | 1 | 1 | 2
  Black or African American | 0 | 0 | 0
  White | 57 | 27 | 84
  Unknown or not reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Summary of Patients Reporting Treatment-Emergent Adverse Events
Description: Overall safety summary of patients experiencing Adverse Events (AEs), Serious Adverse Events (SAEs), treatment-related AEs, and Infusion Associated Reactions (IARs). Summary is based on Treatment-emergent AEs (TEAEs), defined as AEs that occurred following the initiation of study treatment, i.e., alglucosidase alfa or placebo.
Time Frame: weeks 0-78
Population: All patients who received any amount of study treatment comprise the safety population. Patients were considered, for safety analysis, to be in the treatment group of the treatment they actually received.
  Missing or invalid safety or resource utilization data were not replaced.
Measure: Number; unit: participants
Arm/Group | Alglucosidase Alfa | Placebo
Number analyzed (Participants) | 60 | 30
participants
  Patients with Any AEs | 60 | 30
  Patients with Treatment-Related AEs | 32 | 17
  Patients with Infusion-Associated Reactions | 17 | 7
  Patients with SAEs | 13 | 6
  Patients with Severe AEs | 14 | 10
  Patients who Discontinued Due to AEs (incl death) | 3 | 1
  Patients who Died | 1 | 0

2. Primary Outcome: Mean Distance Walked as Measured by Six-minute Walk Test (6MWT) at Weeks 0 and 78, and Mean Change From Baseline
Description: Mean distance walked gives an indication of functional endurance. The greater the distance, the greater the endurance. Mean values of distance walked in a six-minute walk test are offered for baseline, week 78 (or last available observation), and the mean change from baseline (at week 78 or last available post-baseline observation).
Time Frame: weeks 0, 78
Population: Intent-to-Treat (ITT) population. Last observation carried forward. The last available distance walked for one patient was the Baseline visit; therefore, this patient was excluded from the change from baseline calculation.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Alglucosidase Alfa | Placebo
Number analyzed (Participants) | 60 | 30
meters
  Distance Walked at Baseline | 332.20 (126.69) | 317.93 (132.29)
  Distance Walked at Last Available Observation | 357.85 (141.32) | 313.07 (144.69)
  Change at Last Available Observation from Baseline | 26.08 (64.41) | -4.87 (45.24)
Statistical Analysis 1: Comparison: Alglucosidase Alfa vs Placebo; The difference between alglucosidase alfa and placebo treatment groups in change in distance walked from baseline to last observation was estimated by ANCOVA after adjusting for baseline value and randomization strata; Test type: Superiority or Other; p = 0.0347, ANCOVA — The threshold for determining statistical significance is 0.05. A fixed testing sequence procedure was used to preserve an overall error rate of 5% for the co-primary efficacy endpoints by linking the test of FVC to the result of 6MWT; Difference = 28.12, 95% CI [2.07 to 54.17]

3. Primary Outcome: Percent of Predicted Forced Vital Capacity (FVC)
Description: Forced vital capacity is a standard pulmonary function test used to quantify respiratory muscle weakness. Forced vital capacity (FVC) is the volume of air that can forcibly be blown out after full inspiration in the upright position, measured in liters. Predicted forced vital capacity is based on a formula using sex, age and height of a person, and is an estimate of healthy lung capacity. Percent of predicted FVC = (observed value)/(predicted value) * 100%.
Time Frame: weeks 0, 78
Population: ITT population. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: percent predicted FVC
Arm/Group | Alglucosidase Alfa | Placebo
Number analyzed (Participants) | 60 | 30
percent predicted FVC
  Baseline (week 0) | 55.43 (14.44) | 53.00 (15.66)
  Week 78 (or last observation) | 56.71 (16.30) | 50.70 (14.88)
  Change at Week 78 from Baseline | 1.25 (5.55) | -2.30 (4.33)
Statistical Analysis 1: Comparison: Alglucosidase Alfa vs Placebo; The difference between alglucosidase alfa and placebo treatment groups in change in % predicted FVC from baseline to last observation was estimated by ANCOVA after adjusting for baseline value and randomization strata; Test type: Superiority or Other; p = 0.0055, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Difference = 3.40, 95% CI [1.03 to 5.77]

4. Secondary Outcome: Percent Predicted Proximal Muscle Strength of the Lower Limbs as Measured by Quantitative Muscle Testing (QMT)
Description: Quantitative muscle testing (QMT) is a standardized system to measure muscle force production during maximal voluntary isometric contraction. QMT data were collected directly from sensors into laptop computers. Predicted normal values for QMT are based on a formula using sex, age and body mass index of a person, and is an estimate of healthy muscle force. Percent of predicted QMT = (observed value)/(predicted value) * 100%. The QMT Leg Score is the average of the bilateral means for percent predicted knee flexors and extensors. A value of 100% indicates 'normal' muscle strength.
Time Frame: weeks 0, 78
Population: ITT population. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: percent predicted QMT
Arm/Group | Alglucosidase Alfa | Placebo
Number analyzed (Participants) | 60 | 30
percent predicted QMT
  Baseline (week 0) | 37.69 (18.88) | 32.49 (18.24)
  Week 78 (or last available observation) | 39.05 (21.83) | 30.40 (20.54)
  Change at Week 78 from Baseline | 1.22 (9.88) | -2.08 (5.11)
Statistical Analysis 1: Comparison: Alglucosidase Alfa vs Placebo; The difference between alglucosidase alfa and placebo treatment groups in change in QMT from baseline to last observation was estimated by ANCOVA after adjusting for baseline value and randomization strata; Test type: Superiority or Other; p = 0.1093, ANCOVA — The threshold for determining statistical significance is 0.05. No adjustment for multiple comparison was made for secondary efficacy endpoints; Difference = 3.18, 95% CI [-0.73 to 7.08]

5. Secondary Outcome: Health-related Quality of Life Survey Values Related to Physical Components as Measured by the Medical Outcomes Study (MOS) Short Form-36 Health Survey
Description: The Medical Outcomes Study Short Form (MOS SF)-36 questionnaire consists of 36 items grouped into 8 domains designed to assess generic health-related quality of life in healthy and ill adult populations. Physical Component Scores (PCS) report the four domains of physical functioning, role-physical, bodily pain, and general health. Higher scores are associated with better quality of life. All questions are scored on a scale from 0 to 100, with 100 representing the highest level of functioning possible. The PCS scores are reported.
Time Frame: weeks 0, 78
Population: ITT population. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Alglucosidase Alfa | Placebo
Number analyzed (Participants) | 60 | 30
Units on a scale
  PCS at Baseline (week 0) | 34.33 (8.93) | 34.91 (7.26)
  PCS at Week 78 (or last available observation) | 35.11 (9.84) | 36.47 (9.57)
Statistical Analysis 1: Comparison: Alglucosidase Alfa vs Placebo; The difference between alglucosidase alfa and placebo treatment groups in change in PCS from baseline to last observation was estimated by ANCOVA after adjusting for baseline value and randomization strata; Test type: Superiority or Other; p = 0.8333, ANCOVA — [p-value comment as in outcome 4, analysis 1]; Difference = -0.37, 95% CI [-3.83 to 3.09]

6. Primary Outcome: Recombinant Human Acid Alpha-Glucosidase (rhGAA) Pharmacokinetic Parameters: Area Under the Curve (AUC)
Description: Area under the plasma concentration versus time curve from time zero (pre-dose) to 16 hours after the end of infusion. Blood sample time points were 0 (before the start of the infusion), 1 and 2 hours after the start of infusion, end of the infusion, and then 0.25, 0.5, 1, 2, 3, 4, 8, 12,and 16 hours after the end of the infusion (with a 5-minute window for time-points after the start of infusion). Pooled figures combine the values for the three timeframes.
Time Frame: weeks 0, 12 and 52
Population: The subgroup of patients for whom pharmacokinetic samples were obtained was based on those study sites that could accommodate pharmacokinetic sampling needs.
Measure: Mean (Standard Deviation); unit: ug*h/mL
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 32
ug*h/mL
  Week 0 | 2672.47 (1139.85)
  Week 12 | 2386.76 (555.09)
  Week 52 | 2699.28 (999.97)
  Pooled | 2586.17 (933.28)

7. Primary Outcome: Recombinant Human Acid Alpha-Glucosidase (rhGAA) Pharmacokinetic Parameters: Mean Maximum Plasma Concentration(Cmax)
Description: Maximum plasma concentration observed in blood samples taken at the following time points: 0 (before the start of the infusion), 1 and 2 hours after the start of infusion, end of the infusion, and then 0.25, 0.5, 1, 2, 3, 4, 8, 12,and 16 hours after the end of the infusion (with a 5-minute window for time-points after the start of infusion). Pooled figures combine the values for the three timeframes.
Time Frame: weeks 0, 12, 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 32
ng/mL
  Week 0 | 385237 (105585)
  Week 12 | 349269 (78620)
  Week 52 | 369744 (88203)
  Pooled | 368083 (91721)

8. Primary Outcome: Recombinant Human Acid Alpha-Glucosidase (rhGAA) Pharmacokinetic Parameters: Mean Time to Maximum Plasma Concentration(Tmax)
Description: Time to maximum plasma concentration observed in blood samples taken at the following time points: 0 (before the start of the infusion), 1 and 2 hours after the start of infusion, end of the infusion, and then 0.25, 0.5, 1, 2, 3, 4, 8, 12,and 16 hours after the end of the infusion (with a 5-minute window for time-points after the start of infusion). Pooled figures combine the values for the three timeframes.
Time Frame: weeks 0, 12, 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 32
hours
  Week 0 | 3.62 (0.33)
  Week 12 | 3.62 (0.28)
  Week 52 | 3.64 (0.31)
  Pooled | 3.63 (0.30)

ADVERSE EVENTS:
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables. Events are listed independent of relationship to treatment reported.
Arm/Group | Alglucosidase Alfa | Placebo | Overall
Serious Adverse Events (participants affected / at risk) | 13/60 | 6/30 | 19/90
Other Adverse Events (participants affected / at risk) | 60/60 | 30/30 | 90/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alglucosidase Alfa (N=60) | Placebo (N=30) | Overall (N=90)
Coronary artery disease (Cardiac disorders) | 1 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Chest discomfort (General disorders) | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 1
Hypersensitivity (Immune system disorders) | 2 | 0 | 2
Diverticulitis (Infections and infestations) | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Brain stem ischaemia (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Angioneurotic oedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Septal panniculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Aneurysm (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alglucosidase Alfa (N=60) | Placebo (N=30) | Overall (N=90)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 5 | 0 | 5
Macrocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 1
Bundle branch block left (Cardiac disorders) | 1 | 0 | 1
Bundle branch block right (Cardiac disorders) | 1 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 1
Palpitations (Cardiac disorders) | 3 | 1 | 4
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0 | 1
Auricular swelling (Ear and labyrinth disorders) | 1 | 0 | 1
Ear congestion (Ear and labyrinth disorders) | 1 | 1 | 2
Ear discomfort (Ear and labyrinth disorders) | 4 | 1 | 5
Ear pain (Ear and labyrinth disorders) | 3 | 1 | 4
Hypoacusis (Ear and labyrinth disorders) | 20 | 7 | 27
Presbyacusis (Ear and labyrinth disorders) | 1 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 2 | 1 | 3
Tympanic membrane disorder (Ear and labyrinth disorders) | 0 | 1 | 1
Tympanic membrane scarring (Ear and labyrinth disorders) | 0 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 4 | 0 | 4
Altered visual depth perception (Eye disorders) | 1 | 0 | 1
Asthenopia (Eye disorders) | 1 | 0 | 1
Cataract (Eye disorders) | 4 | 2 | 6
Conjunctivitis (Eye disorders) | 1 | 0 | 1
Diplopia (Eye disorders) | 1 | 0 | 1
Dry eye (Eye disorders) | 1 | 0 | 1
Eye irritation (Eye disorders) | 1 | 0 | 1
Eye pruritus (Eye disorders) | 1 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 1 | 1
Photophobia (Eye disorders) | 1 | 0 | 1
Vision blurred (Eye disorders) | 3 | 0 | 3
Visual disturbance (Eye disorders) | 1 | 0 | 1
Vitreous floaters (Eye disorders) | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 2 | 4
Abdominal distension (Gastrointestinal disorders) | 1 | 2 | 3
Abdominal mass (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 3 | 7
Abdominal pain lower (Gastrointestinal disorders) | 2 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 6 | 2 | 8
Constipation (Gastrointestinal disorders) | 6 | 0 | 6
Dental caries (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 18 | 13 | 31
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 5 | 0 | 5
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 2 | 0 | 2
Food poisoning (Gastrointestinal disorders) | 2 | 0 | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 2
Glossodynia (Gastrointestinal disorders) | 0 | 1 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 1
Lip swelling (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 11 | 10 | 21
Oesophageal pain (Gastrointestinal disorders) | 1 | 0 | 1
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 2 | 2
Oral pruritus (Gastrointestinal disorders) | 1 | 0 | 1
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0 | 1
Retching (Gastrointestinal disorders) | 1 | 0 | 1
Stomach discomfort (Gastrointestinal disorders) | 1 | 1 | 2
Swollen tongue (Gastrointestinal disorders) | 2 | 0 | 2
Toothache (Gastrointestinal disorders) | 1 | 4 | 5
Vomiting (Gastrointestinal disorders) | 13 | 3 | 16
Application site vesicles (General disorders) | 1 | 0 | 1
Asthenia (General disorders) | 3 | 4 | 7
Axillary pain (General disorders) | 1 | 0 | 1
Catheter related complication (General disorders) | 1 | 0 | 1
Catheter site pain (General disorders) | 2 | 0 | 2
Catheter site related reaction (General disorders) | 0 | 1 | 1
Chest discomfort (General disorders) | 6 | 1 | 7
Chest pain (General disorders) | 4 | 1 | 5
Chills (General disorders) | 3 | 1 | 4
Fatigue (General disorders) | 7 | 6 | 13
Feeling abnormal (General disorders) | 1 | 0 | 1
Feeling cold (General disorders) | 2 | 0 | 2
Feeling hot (General disorders) | 3 | 2 | 5
Feeling hot and cold (General disorders) | 0 | 1 | 1
Gait disturbance (General disorders) | 1 | 0 | 1
Hangover (General disorders) | 0 | 1 | 1
Influenza like illness (General disorders) | 2 | 4 | 6
Infusion site bruising (General disorders) | 1 | 0 | 1
Infusion site pain (General disorders) | 2 | 0 | 2
Infusion site paraesthesia (General disorders) | 1 | 0 | 1
Infusion site reaction (General disorders) | 5 | 0 | 5
Injection site phlebitis (General disorders) | 1 | 0 | 1
Local swelling (General disorders) | 2 | 1 | 3
Malaise (General disorders) | 3 | 0 | 3
Non-cardiac chest pain (General disorders) | 0 | 1 | 1
Oedema peripheral (General disorders) | 10 | 3 | 13
Pain (General disorders) | 5 | 1 | 6
Pitting oedema (General disorders) | 2 | 2 | 4
Puncture site haemorrhage (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 8 | 8 | 16
Thirst (General disorders) | 1 | 0 | 1
Vessel puncture site haematoma (General disorders) | 0 | 1 | 1
Hypersensitivity (Immune system disorders) | 2 | 0 | 2
Bronchitis (Infections and infestations) | 2 | 1 | 3
Bronchopneumonia (Infections and infestations) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 1
Cystitis (Infections and infestations) | 1 | 1 | 2
Dermatophytosis (Infections and infestations) | 1 | 0 | 1
Eye infection (Infections and infestations) | 1 | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0 | 1
Fungal infection (Infections and infestations) | 1 | 0 | 1
Fungal skin infection (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 5 | 1 | 6
Gastroenteritis viral (Infections and infestations) | 3 | 3 | 6
Gastrointestinal infection (Infections and infestations) | 0 | 2 | 2
Genital infection (Infections and infestations) | 0 | 1 | 1
Gingival infection (Infections and infestations) | 1 | 0 | 1
Herpes simplex (Infections and infestations) | 4 | 3 | 7
Herpes virus infection (Infections and infestations) | 1 | 0 | 1
Influenza (Infections and infestations) | 5 | 7 | 12
Kidney infection (Infections and infestations) | 1 | 1 | 2
Laryngitis (Infections and infestations) | 1 | 0 | 1
Localised infection (Infections and infestations) | 1 | 1 | 2
Mucosal infection (Infections and infestations) | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 25 | 16 | 41
Otitis media (Infections and infestations) | 1 | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0 | 1
Rash pustular (Infections and infestations) | 0 | 1 | 1
Respiratory tract infection (Infections and infestations) | 3 | 0 | 3
Rhinitis (Infections and infestations) | 0 | 2 | 2
Sinusitis (Infections and infestations) | 4 | 4 | 8
Tinea pedis (Infections and infestations) | 2 | 0 | 2
Tonsillitis (Infections and infestations) | 0 | 1 | 1
Tooth infection (Infections and infestations) | 2 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 11 | 3 | 14
Urinary tract infection (Infections and infestations) | 5 | 4 | 9
Vaginal infection (Infections and infestations) | 1 | 0 | 1
Viral infection (Infections and infestations) | 2 | 2 | 4
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 1
Wound infection (Infections and infestations) | 1 | 0 | 1
Accident (Injury, poisoning and procedural complications) | 0 | 1 | 1
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 1 | 2
Back injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 4 | 6 | 10
Excoriation (Injury, poisoning and procedural complications) | 0 | 3 | 3
Fall (Injury, poisoning and procedural complications) | 39 | 20 | 59
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2
Injury (Injury, poisoning and procedural complications) | 4 | 1 | 5
Injury corneal (Injury, poisoning and procedural complications) | 1 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 2 | 3
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 1
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Limb crushing injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 4 | 4 | 8
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 9 | 3 | 12
Repetitive strain injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1 | 2
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 4 | 1 | 5
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 2 | 1 | 3
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Traumatic ulcer (Injury, poisoning and procedural complications) | 1 | 0 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 1 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 2 | 0 | 2
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1
Blood creatine phosphokinase MB increased (Investigations) | 0 | 1 | 1
Blood folate decreased (Investigations) | 1 | 0 | 1
Blood glucose increased (Investigations) | 1 | 1 | 2
Blood parathyroid hormone increased (Investigations) | 0 | 1 | 1
Blood pressure increased (Investigations) | 3 | 1 | 4
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1 | 1
Blood uric acid increased (Investigations) | 1 | 0 | 1
Blood urine present (Investigations) | 1 | 0 | 1
Carbon dioxide increased (Investigations) | 0 | 1 | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 | 1 | 2
Eosinophil count increased (Investigations) | 0 | 1 | 1
Forced expiratory volume decreased (Investigations) | 0 | 1 | 1
Glucose urine present (Investigations) | 1 | 0 | 1
Heart rate irregular (Investigations) | 0 | 1 | 1
International normalised ratio decreased (Investigations) | 0 | 1 | 1
Lymph node palpable (Investigations) | 0 | 1 | 1
Neutrophil count increased (Investigations) | 1 | 0 | 1
Oxygen saturation decreased (Investigations) | 1 | 0 | 1
Protein total increased (Investigations) | 0 | 1 | 1
Protein urine present (Investigations) | 1 | 0 | 1
Specific gravity urine decreased (Investigations) | 0 | 1 | 1
Urine ketone body present (Investigations) | 1 | 0 | 1
Vitamin D decreased (Investigations) | 0 | 1 | 1
Weight decreased (Investigations) | 2 | 0 | 2
Weight increased (Investigations) | 0 | 1 | 1
White blood cell count increased (Investigations) | 1 | 0 | 1
White blood cells urine positive (Investigations) | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1
Diabetes mellitus non-insulin-dependent (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 9 | 27
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 7 | 21
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 14 | 6 | 20
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Muscle twitching (Musculoskeletal and connective tissue disorders) | 5 | 1 | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 | 3 | 9
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 | 1 | 6
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 | 2 | 10
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 8 | 1 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 5 | 17
Neck pain (Musculoskeletal and connective tissue disorders) | 7 | 5 | 12
Nose deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 | 7 | 22
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Areflexia (Nervous system disorders) | 3 | 2 | 5
Balance disorder (Nervous system disorders) | 0 | 1 | 1
Burning sensation (Nervous system disorders) | 2 | 0 | 2
Carpal tunnel syndrome (Nervous system disorders) | 1 | 1 | 2
Disturbance in attention (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 14 | 6 | 20
Dizziness postural (Nervous system disorders) | 2 | 0 | 2
Dysgeusia (Nervous system disorders) | 0 | 1 | 1
Facial palsy (Nervous system disorders) | 1 | 0 | 1
Head discomfort (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 24 | 15 | 39
Hyperreflexia (Nervous system disorders) | 1 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 2 | 2 | 4
Hyporeflexia (Nervous system disorders) | 2 | 1 | 3
Intercostal neuralgia (Nervous system disorders) | 1 | 0 | 1
Intracranial hypotension (Nervous system disorders) | 0 | 1 | 1
Lethargy (Nervous system disorders) | 2 | 0 | 2
Loss of consciousness (Nervous system disorders) | 2 | 0 | 2
Migraine (Nervous system disorders) | 3 | 1 | 4
Nerve compression (Nervous system disorders) | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 6 | 4 | 10
Poor quality sleep (Nervous system disorders) | 0 | 1 | 1
Sinus headache (Nervous system disorders) | 1 | 1 | 2
Somnolence (Nervous system disorders) | 3 | 0 | 3
Syncope vasovagal (Nervous system disorders) | 1 | 1 | 2
Tremor (Nervous system disorders) | 4 | 0 | 4
Abnormal dreams (Psychiatric disorders) | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 2 | 3 | 5
Depression (Psychiatric disorders) | 1 | 2 | 3
Insomnia (Psychiatric disorders) | 6 | 2 | 8
Panic attack (Psychiatric disorders) | 0 | 1 | 1
Stress (Psychiatric disorders) | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 3 | 1 | 4
Leukocyturia (Renal and urinary disorders) | 1 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 3 | 0 | 3
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 1
Proteinuria (Renal and urinary disorders) | 2 | 1 | 3
Pyuria (Renal and urinary disorders) | 1 | 2 | 3
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 1
Urine flow decreased (Renal and urinary disorders) | 1 | 0 | 1
Urine odour abnormal (Renal and urinary disorders) | 1 | 1 | 2
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 1
Breast swelling (Reproductive system and breast disorders) | 1 | 0 | 1
Breast tenderness (Reproductive system and breast disorders) | 1 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 2 | 2
Fibrocystic breast disease (Reproductive system and breast disorders) | 1 | 0 | 1
Genital pruritus female (Reproductive system and breast disorders) | 0 | 1 | 1
Menstrual discomfort (Reproductive system and breast disorders) | 1 | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 1 | 1 | 2
Scrotal cyst (Reproductive system and breast disorders) | 0 | 1 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 11
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 | 5 | 17
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 5
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Erythema (Skin and subcutaneous tissue disorders) | 3 | 1 | 4
Heat rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 | 0 | 5
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 1 | 7
Rash (Skin and subcutaneous tissue disorders) | 6 | 3 | 9
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 3 | 0 | 3
Rash pruritic (Skin and subcutaneous tissue disorders) | 4 | 1 | 5
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Skin nodule (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin warm (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 6 | 0 | 6
Aneurysm (Vascular disorders) | 1 | 0 | 1
Diastolic hypotension (Vascular disorders) | 1 | 0 | 1
Flushing (Vascular disorders) | 3 | 2 | 5
Haematoma (Vascular disorders) | 2 | 0 | 2
Hot flush (Vascular disorders) | 1 | 1 | 2
Hypertension (Vascular disorders) | 3 | 1 | 4
Hypotension (Vascular disorders) | 2 | 1 | 3
Phlebitis (Vascular disorders) | 0 | 1 | 1
Raynaud's phenomenon (Vascular disorders) | 1 | 1 | 2
Vasoconstriction (Vascular disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, PI can publish after Genzyme publishes or 18 months after study completion. PI gives Genzyme a draft 60 days before publication. Genzyme can ask that confidential information be removed, and can defer publication another 60 days upon notifying PI that it will file a patent application on inventions contained in the draft.